CLINICAL TRIAL: NCT06764992
Title: Exploring Men s Prostate Cancer Genetic Risk Perceptions and Willingness to Give a Biospecimen for Genetic Risk Testing
Brief Title: Exploring Men s Prostate Cancer Genetic Risk Perceptions
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-21876
Record Dates: First submitted 2025-01-07; First posted 2025-01-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Genetic Risk Perception and Beliefs; Biospecimen Donation for Genetic Risk Testing
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to provide a saliva sample. Each enrolled participant will be provided the Oragene saliva collection kit (opt in) with collection, storage and mailing instructions per established protocols DNA extraction and genotyping assay will be done in Dr. Park's (PI) laboratory and Moffitt Cancer Center's Molecular Genomic Core facility, respectively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer Risk Group: Participants will be asked to provide saliva samples and complete a questionnaire about their Prostate Cancer Genetic Risk beliefs.
  Interventions: Other: Questionnaire; Other: Saliva Sample

INTERVENTIONS:
Other: Questionnaire — Participants will be asked to complete a questionnaire on demographics, risk beliefs and perception and prostate cancer screening behaviors, intentions and awareness of informed decision making.
Other: Saliva Sample — Participants will be asked to provide a saliva sample for genetic risk testing to generate a SNP risk profile using a saliva sample collection kit with collection, storage and mailing instructions. We will assess the proportion of consented men who will provide a saliva sample.

SUMMARY:
The exploring men's prostate cancer genetic risk perceptions and willingness to give a biospecimen for genetic risk testing study aims to assess prostate cancer genetic risk and susceptibility beliefs among unaffected men of diverse races/ethnicities who are considering undergoing prostate cancer screening and their willingness of men to provide a biospecimen (saliva sample) and test the samples for prostate cancer aggressiveness and determine risk category based on SNP genetic profile.

ELIGIBILITY:
Inclusion Criteria:

* Racially/ethnically diverse men with emphasis on Men of African Ancestry.
* Age 40 and older .
* No personal prostate cancer history/diagnosis.
* With or without family history of prostate cancer.

Exclusion Criteria:

* Previous personal Prostate Cancer history/diagnosis
* Under 40 years of age

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This Study is evaluating Prostate Cancer risk
Study Population: Racially and ethnically diverse Adult Men with no personal Prostate Cancer history/diagnosis.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Prostate Cancer Genetic Risk and Susceptibility Beliefs | Up to 6 Months
  Prostate Cancer Genetic Risk and Susceptibility beliefs will be summarized based on single items on the Prostate Cancer Risk Perception Questionnaire.

SECONDARY OUTCOMES:
Polygenic Risk Score (PRS) of Saliva Samples | Up to 6 Months
  Polygenic Risk Score (PRS) of Saliva Samples will be based on genetic profiles from Single Nucleotide Polymorphisms (SNPs).
  Identified as prostate cancer susceptibility loci, genetic risk of developing prostate cancer will be categorized into 5 groups:
  Very Low Risk (< 10%), Low Risk (10-25%) Moderate Risk (25-75%), High Risk (75-90%) or Very High Risk (>90%).

CONTACTS AND LOCATIONS:
Overall Officials: Jong Park, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/